CLINICAL TRIAL: NCT01591603
Title: Comparison of Perineural Catheter Depth for the Continuous Popliteal Nerve Block Using Ultrasound Guidance and Dermabond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Clifford Bowens, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120382
Record Dates: First submitted 2012-04-23; First posted 2012-05-04 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Neuromuscular Inhibition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Procedure: 1 cm
- Group 2 (Experimental)
  Interventions: Procedure: 5 cm

INTERVENTIONS:
Procedure: 1 cm — A Tuohy needle will be advanced in-plane with the bevel cephalad to a point that lies between the tibial and common peroneal branches of the sciatic nerve. The catheter will be advanced 1 cm past the tip of the Tuohy
  Other Names: 18 gauge 100mm Contiplex Tuohy needle; 20-gauge non-stimulating catheter
  Arms: Group 1
Procedure: 5 cm — A Tuohy needle will be advanced in-plane with the bevel cephalad to a point that lies between the tibial and common peroneal branches of the sciatic nerve. The catheter will be advanced 5 cm past the tip of the Tuohy
  Other Names: 18 gauge 100mm Contiplex Tuohy needle; 20-gauge non-stimulating catheter
  Arms: Group 2

SUMMARY:
The study will investigate the difference in success rate between popliteal peripheral nerve catheters placed at 1 centimeter compared to 5 centimeters past the tip of a Tuohy needle.

DETAILED DESCRIPTION:
Traditionally for the lower extremity, peripheral nerve catheters have been threaded greater than or equal to 5 centimeters past the tip of the Tuohy needle. The major rational for this practice is to reduce dislodgement. However, the greater the distance that a catheter is advanced, the greater the risk of contacting undesired structures, kinking, looping and knotting. For the continuous popliteal nerve block, the catheter is threaded perpendicular to the course of the nerve. This could result in the tip of the catheter being a significant distance from the targeted nerve which may lead to a decrease in the success rate or efficacy of the block.

Greater efficacy may be seen if the needle is closer to its target. This may be quantified by documenting a faster onset of motor and sensory changes and/or a lower catheter infusion rate required to maintain pain control. The study will investigate the difference in success rate between popliteal peripheral nerve catheters placed at 1 centimeter compared to 5 centimeters past the tip of a Tuohy needle.

ELIGIBILITY:
Inclusion Criteria:

* Will be having a popliteal nerve blocks
* Do not meet any of the exclusion criteria listed below.

Exclusion Criteria:

* < 18 years old
* BMI > 35
* Pregnant patients
* Diabetes mellitus or patients with known neuropathy
* Amputations & polytrauma patients
* Patients allergic to local anesthetics
* Chronic Pain patients
* Patients in whom communication is a problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Peripheral block score (PBS). | 10, 20, and 30 minutes after intervention
  The extent of popliteal nerve blockade will be captured with four sensory groups (sural, superficial peroneal, tibial, and deep peroneal) and three motor groups (superficial peroneal, tibial, and deep peroneal). For each group, a score of 0, 1, or 2 will be assigned based on complete, partial, or no blockade, respectively. The peripheral block score (PBS) outcome variable will be based on the sum of these values and will range from 0 to 14.

SECONDARY OUTCOMES:
Pain score | Arrival to PACU (Immediately after surgery, approximately 3-5 hours after intervention)
  The investigators will examine the difference in the pain scores (0-10 numeric rating scale) between the two groups.
Analgesia failure rate | Arrival to PACU (Immediately after surgery, approximately 3-5 hours after intervention)
  The investigators will examine the difference in analgesia failure rates in the PACU. Analgesia failure is defined as the failure of a rescue bolus (to treat patient pain).
Catheter dislodgement rates | Arrival to PACU (Immediately after surgery, approximately 3-5 hours after intervention)
  The investigators will examine the difference in the catheter dislodgement rates.
Difference in total opioid usage | Length of Stay In PACU (Approximately 5-7 hours after intervention)
  The investigators will examine the difference in the total opioid usage. We will compare medications separately and in total equivalent units (using an opioid conversion table).
Degree of Doppler color agitation | Immediately after intervention
  The investigators will examine the relationship between the degree of Doppler color agitation (evaluated at the time the catheter is placed) and block success (i.e., the outcome in the primary analysis). Degree of agitation color will be defined as the percentage of nerve covered during the color agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Bowens, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Bowens C Jr, Badiola IJ, Allen BFS, Canlas CL, Gupta RK, Jaeger LM, Briggs ER, Corey JM, Shi Y, Schildcrout JS, Malchow RJ. Color Doppler ultrasonography of an agitated solution is predictive of accurate catheter placement for a continuous popliteal sciatic nerve block. Perioper Med (Lond). 2021 Dec 15;10(1):59. doi: 10.1186/s13741-021-00229-w. PMID 34906248